CLINICAL TRIAL: NCT00726843
Title: Evaluation of Yoga for the Treatment of Pediatric Headaches
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Enrollment proceeded too slowly to conduct study as RCT.
Sponsor: Medical College of Wisconsin (Other)
Collaborators: Children's Hospital and Health System Foundation, Wisconsin (Other); Santosh Yoga LLC (Industry)
Responsible Party: Principal Investigator, Keri Hainsworth, Associate Professor, Medical College of Wisconsin
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 85067-3
Record Dates: First submitted 2008-07-30; First posted 2008-08-01 (Estimated); Last update posted 2015-04-07 (Estimated); Status verified 2015-04

CONDITIONS: Headache
Keywords: Headache; Complementary and Alternative Medicine; Pediatric; Yoga
MeSH Terms: conditions — Headache

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Active Comparator): 8 weeks of Yoga, followed by 8 weeks of follow-up
  Interventions: Other: 8 weeks of Iyengar Yoga
- 2 (Active Comparator): 8 weeks of follow-up, followed by 8 weeks of yoga
  Interventions: Other: 8 weeks of Iyengar Yoga

INTERVENTIONS:
Other: 8 weeks of Iyengar Yoga — Participants will attend 8 weekly, 75 min. yoga sessions, followed by 8 weeks of follow-up (will provide headache frequency/intensity)
  Arms: 1
Other: 8 weeks of Iyengar Yoga — Participants will provide headache frequency/intensity for 8 weeks, followed by 8 weekly, 75 min. yoga sessions
  Arms: 2

SUMMARY:
This study will examine the feasibility and acceptability of yoga for adolescents seen by a medical practitioner for their headaches. The study will also examine whether yoga decreases anxiety and improves quality of life. We hypothesize that yoga will be both acceptable and feasible with a pediatric population. We also hypothesize that yoga will decrease anxiety and improve quality of life.

ELIGIBILITY:
Inclusion Criteria:

* 13-17 years
* patient seen in the headache clinic at Children's Hospital of Wisconsin

Exclusion Criteria:

* neck, spinal, or back injuries

Ages: 13 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 7 (Actual)
Dates: Start 2008-07; Primary Completion 2008-12 (Actual); Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
Headache Pain | Pre; Post; Weekly

SECONDARY OUTCOMES:
Yoga Attendance | weekly

CONTACTS AND LOCATIONS:
Overall Officials: Keri R Hainsworth, Ph.D., Principal Investigator — Medical College of Wisconsin
Locations (1):
- Children's Hospital of Wisconsin, Milwaukee, Wisconsin, United States